CLINICAL TRIAL: NCT05050955
Title: AlloSure Lung Assessment and Metagenomics Outcomes Study
Acronym: ALAMO
Status: Active, not recruiting | Type: Observational
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-C-00016
Record Dates: First submitted 2021-08-30; First posted 2021-09-21 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Lung Transplant Infection; Lung Transplant; Complications; Lung Transplant Failure and Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LungCare Surveillance (500 Cases): Observational evaluation of diagnostic performance characteristics of AlloSure Lung to detect a spectrum of rejection and allograft infection.

SUMMARY:
ALAMO is a prospective, multi-center, perspective, registry of patients receiving LungCare™ (AlloSure®-Lung, AlloMap Lung, and HistoMap) for surveillance post-transplant. This study aims to evaluate the diagnostic performance characteristics of AlloSure Lung (dd-cfDNA) to detect a spectrum of rejection (ACR, AMR) and allograft infection (Bacterial, Viral, Fungal, Mycobacterial, Parasitic).

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational registry of lung transplant recipients receiving LungCare (AlloSure-Lung, AlloMap Lung, and Histomap) surveillance testing. Patients will be recruited based on utilization of surveillance testing with LungCare, as deemed appropriate for their care post-transplant. Patients deemed eligible for the study by their physician will be invited to participate during their usual care visit. Enrolled patients will receive evaluations and treatment for their lung transplant according to their health care provider and clinical practice at each study site. Treatment and follow-up visits will be determined by the treating physician. Information related to surveillance testing, selected clinical outcomes, and treatments received for managing the lung transplant recipients will be collected from medical records. The product Laboratory Services Guide(s) will be provided as a reference. Patient data (including diagnosis and biopsy outcomes) will be drawn from the patients' medical records. This data will be recorded by the site study personnel via a web-based electronic data collection (EDC) system every month.

The study is designed to observe the clinical use of LungCare and patient outcomes in a cohort of lung transplant recipients managed with LungCare. This cohort design is selected because it is efficient and effective to evaluate the real-world robust performance of LungCare on patient management and outcomes that can be generalized to the intended use population. A well-designed observational cohort study that includes a large number of patients with long-term follow-up may provide robust results with several advantages, such as gathering data regarding sequence of events to assess causality; examining multiple outcomes for a given LungCare use; calculating rates of biopsy and rejection; and operational efficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral or Bilateral, deceased-donor, initial or re-transplant
2. ≤ 90 days post-transplant
3. Ability to understand and provide informed consent and adhere to laboratory surveillance schedule
4. Patients who have LungCare initiated within 30 days of signing the informed consent form

Exclusion Criteria:

1. Multi-organ transplants
2. Pregnancy
3. Active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All lung transplant patients without exclusion criteria will be eligible to enter the study. Patients will be approached by the study team at the time of listing or at the time of transplant or within 90 days post-transplant to discuss the trial, consent and enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
ALAD | 1 year post-transplant
  Diagnostic performance characteristics (sensitivity, specificity, PPV, NPV) of AlloSure Lung to detect acute lung allograft dysfunction (ALAD).

SECONDARY OUTCOMES:
Chronic lung allograft dysfunction | 3 years post-transplant
  Clinical diagnostic performance characteristics (sensitivity, specificity, PPV and NPV) of AlloSure Lung to detect chronic lung allograft dysfunction.
Acute cellular rejection | 3 years post-transplant
  Clinical diagnostic performance characteristics (sensitivity, specificity, PPV and NPV) of AlloSure Lung to detect acute cellular rejection (ACR).
Antibody mediated rejection | 3 years post-transplant
  Clinical diagnostic performance characteristics (sensitivity, specificity, PPV and NPV) of AlloSure Lung to detect antibody mediated rejection (AMR).
Acute infection | 3 years post-transplant
  Clinical diagnostic performance characteristics (sensitivity, specificity, PPV and NPV) of AlloSure Lung to detect acute infection.
Subject Variability | 3 years post-transplant
  Define within-subject and between-subject variability of AlloSure Lung in clinically stable patients in order to establish reference change value RCV.
ALAD vs. Stability | 3 years post-transplant
  Evaluate the diagnostic performance characteristics of utilizing RCV to distinguish ALAD vs. Stability
Biopsy-proven rejections | 3 years post-transplant
  The proportion of biopsy-proven rejections with elevated AlloSure Lung versus those without elevated AlloSure-Lung.
AlloSure Lung Results | 3 years post-transplant
  The proportion of AlloSure Lung results obtained as surveillance or for-cause, that the physicians felt influenced their decisions around management of patients.
ALAD Free survival | 3 years post-transplant
  ALAD free survival in lung transplant recipients who received AlloSure Lung as part of post-transplant surveillance.
AlloSure Levels | 3 years post-transplant
  Evaluate AlloSure levels 30-90 days prior to acute rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Levine, Principal Investigator — Stanford University; Nirmal Sharma, Principal Investigator — Brigham and Women's Hospital
Locations (22):
- United States (21):
  - University of Alabama (UAB), Birmingham, Alabama
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California (UCSF) School of Medicine, San Francisco, California
  - University of CO Anschutz Medical Campus, Aurora, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - Loyola University Medical School, Maywood, Illinois
  - University of Louisville Health, Louisville, Kentucky
  - University of Mayland, Baltimore, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Washington University-Barnes Jewish Hospital, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Health/ Memorial Hermann Hospital, Houston, Texas
  - Inova, Falls Church, Virginia
  - University of Wisconsin Madison, Madison, Wisconsin
- Toronto General Hospital, Toronto, Ontario, Canada